CLINICAL TRIAL: NCT05270863
Title: Multicenter, Double-Masked, Randomized, Safety and Efficacy Study of BRIMOCHOL™ PF and Carbachol PF Topical Ophthalmic Solution With Emmetropic Phakic and Pseudophakic Presbyopia
Brief Title: Safety and Efficacy Study BRIMOCHOL™ PF and Carbachol PF in Subjects With Emmetropic Phakic or Pseudophakic Presbyopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Visus Therapeutics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VT-002
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Carbachol; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BRIMOCHOL™ PF (Experimental): A single drop in each eye at a visit.
  Interventions: Drug: BRIMOCHOL™ PF
- Carbachol PF (Active Comparator): A single drop in each eye at a visit.
  Interventions: Drug: Carbachol PF
- Brimonidine tartrate (Active Comparator): A single drop in each eye at a visit.
  Interventions: Drug: Brimonidine tartrate

INTERVENTIONS:
Drug: BRIMOCHOL™ PF — A single drop in each eye at a visit.
  Other Names: carbachol/brimonidine tartrate
  Arms: BRIMOCHOL™ PF
Drug: Carbachol PF — A single drop in each eye at a visit.
  Other Names: carbachol monotherapy
  Arms: Carbachol PF
Drug: Brimonidine tartrate — A single drop in each eye at a visit.
  Other Names: brimonidine tartrate monotherapy
  Arms: Brimonidine tartrate

SUMMARY:
Safety and Efficacy Study of BRIMOCHOL™ PF and Carbachol PF in Subjects With Emmetropic Phakic and Pseudophakic Presbyopia

DETAILED DESCRIPTION:
Multicenter, Double-Masked, Randomized, Safety and Efficacy Study of BRIMOCHOL™ PF and Carbachol PF Topical Ophthalmic Solution With Emmetropic Phakic and Pseudophakic Presbyopia

ELIGIBILITY:
Inclusion Criteria:

* Male or female in good general health
* Must have presbyopia

Exclusion Criteria:

* History of allergic reaction to the study drug or any of its components
* Any disease or medical condition that, in the opinion of the Investigator, would prevent the subject from participating in the study or might confound study results

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Visus Therapeutics Investigative Site, Glendale, California
  - Visus Therapeutics Investigative Site, Rancho Cordova, California
  - Visus Therapeutics Investigative Site, Jacksonville, Florida
  - Visus Therapeutics Investigative Site, Morrow, Georgia
  - Visus Therapeutics Investigative Site, Roswell, Georgia
  - Visus Therapeutics Investigative Site, Shawnee Mission, Kansas
  - Visus Therapeutics Investigative Site, Kansas City, Missouri
  - Visus Therapeutics Investigative Site, Pittsburgh, Pennsylvania
  - Visus Therapeutics Investigative Site, Memphis, Tennessee
  - Visus Therapeutics Investigative Site, Cedar Park, Texas
  - Visus Therapeutics Investigative Site, Houston, Texas
  - Visus Therapeutics Investigative Site, San Antonio, Texas
  - Visus Therapeutics Investigative Site, Ogden, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B, C, BF: Crossover design with 3 study treatments. Participants received Brimonidine, Carbachol PF, or BRIMOCHOL PF.
- B, BF, C: Crossover design with 3 study treatments. Participants received Brimonidine, BRIMOCHOL PF, or Carbachol PF.
- C, B, BF: Crossover design with 3 study treatments. Participants received Carbachol PF, Brimonidine, or BRIMOCHOL PF.
- C, BF, B: Crossover design with 3 study treatments. Participants received Carbachol PF, BRIMOCHOL PF, or Brimonidine
- BF, B, C: Crossover design with 3 study treatments. Participants received BRIMOCHOL PF, Brimonidine, or Carbachol PF.
- BF, C, B: Crossover design with 3 study treatments. Participants received BRIMOCHOL PF, Carbachol PF, or Brimonidine.
Period: Visit 2 First Intervention
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 31 | 30 | 30 | 30 | 31 | 30
Completed | 31 | 30 | 30 | 29 | 31 | 30
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Randomization error | 0 | 0 | 0 | 1 | 0 | 0
Period: First Washout
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 31 | 30 | 30 | 29 | 31 | 30
Completed | 31 | 30 | 30 | 29 | 30 | 28
Not Completed | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Period: Visit 3 Second Intervention
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 31 | 30 | 30 | 29 | 30 | 28
Completed | 30 | 30 | 29 | 29 | 30 | 28
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Inclusion Criteria | 1 | 0 | 1 | 0 | 0 | 0
Period: Second Washout
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 30 | 30 | 29 | 29 | 30 | 28
Completed | 29 | 29 | 29 | 28 | 30 | 28
Not Completed | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Period: Visit 4 Third Invervention
Arm/Group | B, C, BF | B, BF, C | C, B, BF | C, BF, B | BF, B, C | BF, C, B
Started | 29 | 29 | 29 | 28 | 30 | 28
Completed | 29 | 29 | 29 | 28 | 30 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: 3 study treatments across 4 study visits
Arm/Group | All Subjects
Number analyzed (Participants) | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47
  Not Hispanic or Latino | 135
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 46
  White | 116
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 182

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With >=15 Letter Gain Without >=5 Letter Loss in Near Visual Acuity
Description: Primary endpoint measure at hour 1 post-dose at study visit
Time Frame: Day 1 Hour 1
Population: All participants who received at least one dose of study treatment (mITT)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BRIMOCHOL™ PF | Carbachol PF | Brimonidine Tartrate
Number analyzed (Participants) | 178 | 177 | 176
Percentage of participants | 49.4 [41.9 to 57.0] | 35.0 [28.0 to 42.5] | 22.7 [16.8 to 29.6]
Statistical Analysis 1: Comparison: BRIMOCHOL™ PF vs Carbachol PF vs Brimonidine Tartrate; Test type: Superiority; p < .001, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 45 Days
Arm/Group | BRIMOCHOL™ PF | Carbachol PF | Brimonidine Tartrate
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/177 | 0/176
Serious Adverse Events (participants affected / at risk) | 1/178 | 0/177 | 0/176
Other Adverse Events (participants affected / at risk) | 37/178 | 24/177 | 2/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRIMOCHOL™ PF (N=178) | Carbachol PF (N=177) | Brimonidine Tartrate (N=176)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BRIMOCHOL™ PF (N=178) | Carbachol PF (N=177) | Brimonidine Tartrate (N=176)
Eye Irritation (Eye disorders) | 25 | 20 | 1
Headache (Nervous system disorders) | 16 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT05270863/Prot_002.pdf
  • Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT05270863/SAP_003.pdf